CLINICAL TRIAL: NCT02535793
Title: Characterisation of Occupational Allergy to Drosophila
Acronym: DROSOALLERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF 9410
Record Dates: First submitted 2015-08-20; First posted 2015-08-31 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Drosophila; Clinical Symptoms
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laboratory workers with symptoms in presence of drosophila (Other)
  Interventions: Other: blood test (four dry tubes 7ml) and prick tests

INTERVENTIONS:
Other: blood test (four dry tubes 7ml) and prick tests

SUMMARY:
Allergy is a very common problem and can be a handicap in everyday life, specially when symptoms occur at work place. Some persons working with drosophila developed respiratory symptoms. Investigators tried to analyze if these manifestations could be due to a specific allergy to drosophila.

DETAILED DESCRIPTION:
To do so, investigators invited laboratory workers who presented any symptoms in presence of drosophila to undergo skin prick tests in order to determine if a specific sensibilization to drosophila exists. Then, a blood sample is taken from these persons to research specific IgE directed against drosophila. By this way, investigators hope determine if a specific allergy to drosophila exists, its characteristics as prevalence, symptoms, populations concerned...in order to better protect laboratory workers and prevent allergy incidence.

ELIGIBILITY:
Inclusion Criteria:

* major males or females (aged <68) who work in laboratory with drosophila in Montpellier (France)
* clinical symptoms in presence of drosophila
* The subject must be affiliated to a social security scheme
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* The patient has indicated against (or incompatible drug combination) concerning the implementation of a prick test
* antihistamine cure in progress
* Inability to understand the nature and goals of the study and / or communication difficulties with the investigator
* No affiliation to a French social security recipient or not such a scheme
* Major protected by law (guardianship, curator or under judicial protection)
* deprivation of liberty by judicial or administrative decision
* Increased likelihood of non compliance to the protocol or abandonment under study
* pregnancy or breastfeeding

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with positive prick test to drosophila | The day of inclusion
  Prick tests : measuring the size of the skin reaction (wheal) after prick tests with drosophila. A wheal measuring more than 4 millimeters in diameter sign a sensitization to drosophila. Then, a blood sample is collected in order to measure specific drosophila IgE rate

SECONDARY OUTCOMES:
Survey to analyse risk factors for allergy to drosophila | The day of inclusion
  analysis of professional (attended institute, time from start working with drosophila, type of animal manipulation (species, living, dead, DNA, protein) use of protection,) or personal factors (age, gender, others allergies, treatment used) which could lead to allergic reaction to drosophila

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Arnaud de Villeneuve, Montpellier, France